CLINICAL TRIAL: NCT05020145
Title: Coronavirus Disease 2019 (COVID-19) Vaccination and Breakthrough Infections Among Persons With Immunocompromising Conditions in the United States
Brief Title: COVID-19 Vaccination and Breakthrough Infections Among Persons With Immunocompromising Conditions in the United States
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591035
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Immunocompromised; Immunosuppressed; Covid-19; SARS-COV-2; SARS-COV-2 Infection; Breakthrough Infection
Keywords: Immunocompromised; Immunosuppressed; Immunosuppressive drugs; Covid-19; Covid-19 Vaccination; mRNA Vaccine; SARS-CoV-2 Vaccine; BNT162b2; Breakthrough Infection; SARS-COV-2 Infection; SARS-COV-2
MeSH Terms: conditions — COVID-19; Breakthrough Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Immunocompromised: Vaccinated Subject with 1 or >1 immunocompromising conditions.
  Interventions: Biological: BNT162b2 (Tozinameran)
- Non-Immunocompromised: Vaccinated subjects without evidence of immunocompromising condition.
  Interventions: Biological: BNT162b2 (Tozinameran)
- Total Population (immunocompromised and non): Vaccinated Subjects with or without 1 or >1 immunocompromising conditions.
  Interventions: Biological: BNT162b2 (Tozinameran)

INTERVENTIONS:
Biological: BNT162b2 (Tozinameran) — Covid-19 Vaccine
  Other Names: Pfizer-BioNTech COVID-19 vaccine

SUMMARY:
This retrospective study will evaluate characteristics, vaccine utilization and outcomes among subjects with immunocompromising conditions that received COVID-19 vaccination.

DETAILED DESCRIPTION:
The objective of this US-based retrospective cohort study is to evaluate characteristics, vaccine utilization and outcomes among subjects with immunocompromising conditions that received COVID-19 vaccination.

Subjects will be aged 12 years and older and will have no evidence of prior SARS-CoV-2 infection.

The primary analysis will be conducted on subjects vaccinated with BNT162b2.

A variety of subgroup analyses and sensitivity analyses are planned.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Unique enrollees in the HealthVerity Vaccine dataset anytime after December 10, 2020
2. At least 12 years on the index date (ie, first vaccination date)
3. No evidence of prior COVID-19 infection (a medical claim, pharmacy claim, or chargemaster record with a diagnosis code of ICD-10-CM U07.1) in the 12 months prior to the index date
4. Have 12 months of continuous enrollment with medical benefits (with or without pharmacy benefits) prior to the index date.

Subjects with an IC condition will be identified via an algorithm developed for use in administrative claims database studies.

Exclusion criteria: subjects not meeting the criteria above will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The main study population consists of subjects >12 that received Covid-19 vaccination, had no evidence of prior infection, had continuous enrollment and evidence of immunocompromising conditions during the baseline pre vaccination period.
Sampling Method: Non-Probability Sample
Enrollment: 1277747 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants aged 12 years or more with at least 1 BNT162b2 vaccine claim between 10 Dec 2020 to 08 Jul 2021 examined for COVID-19 breakthrough infections (vaccination greater than equal to [>=] 14 days after 2nd dose) in real-world practice, were retrieved from US HealthVerity database. Available data were extracted and evaluated during approximately 4 months of this retrospective observational study.
Groups:
- BNT162b2 (Tozinameran): IC Cohort: Participants with IC condition who had at least 1 BNT162b2 vaccine claim between 10 December 2020 to 08 July 2021 were retrospectively observed in this cohort. Participants were considered immunocompromised if they had >=1 hospitalization or >=2 outpatient visits on separate dates on a healthcare claim indicated 1 or more IC condition or if they had usage of specific immunosuppressive (IS) medications during the 12-month baseline period (prior to index period). Index date was defined as the date of receipt of the 1st BNT162b2 dose.
- BNT162b2 (Tozinameran): Non-IC Cohort: Participants who had at least 1 BNT162b2 vaccine claim between 10 December 2020 to 08 July 2021 and without evidence of immunocompromising condition were included in this reporting arm.
Period: Overall Study
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Started | 225796 | 1051951
Fully Vaccinated | 212945 | 963962
Completed | 225796 | 1051951
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants at least 12 years of age with at least one vaccine claim between 10 Dec 2020 to 08 Jul 2021 from the HealthVerity health care database, had 12 months of continuous medical enrollment prior to the receipt of their first vaccine with no evidence of a SARS-CoV-2 infection in the year prior to being vaccinated.
Groups:
- Total: Total of all reporting groups
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort | Total
Number analyzed (Participants) | 225796 | 1051951 | 1277747
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (15.2) | 44.1 (16.9) | 46.1 (17.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 127101 | 558164 | 685265
  Male | 96835 | 476804 | 573639
  Unknown | 1860 | 16983 | 18843
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Breakthrough Cases of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Description: The incidence rate of breakthrough cases of SARS-CoV-2 infection was calculated as the number of participants who experienced the event divided by the observed time at risk and reported as incidence rate per 100 person-years. Rate of breakthrough SARS-CoV-2 infection among fully vaccinated participants was reported in this outcome measure.
Time Frame: From 14 days after Dose 2 of BNT162b2 vaccine up to COVID-19 vaccine breakthrough infection case or end of continuous enrollment, whichever occurred first (retrospective data was retrieved and observed during 4 months approximately)
Population: Analysis population included fully vaccinated participants against COVID-19 in dataset during 10-Dec-2020 through 08-Jul-2021, at least 12 years old on index date, had continuous medical enrolment 12-month period prior to index date, with no prior COVID-19 diagnosis during baseline. Fully vaccinated was defined as >=14 days of follow-up after Dose 2 of BNT162b2 vaccine. Here, N=participant who had at least 1 incidence of SARS-CoV-2 breakthrough infection were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 212945 | 963962
Events per 100 person-years | 0.89 [0.80 to 0.98] | 0.34 [0.32 to 0.37]

2. Primary Outcome: Time to SARS-CoV-2 Breakthrough Infection
Description: Time to SARS-CoV-2 breakthrough infection was calculated as the number of days from Dose 2 of vaccination till first occurrence of a breakthrough SARS-CoV-2 infection.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 374 | 604
Days | 34.5 [22 to 58] | 33 [20.5 to 58]

3. Secondary Outcome: Number of Participants With Emergency Department Visits After SARS-CoV-2 Infection
Description: In this outcome measure, number of participants with emergency department visits who were fully vaccination and had SARS-CoV-2 breakthrough infection were analyzed. Emergency department visits included an outpatient claim that occurs after the breakthrough COVID-19 diagnosis date or at the same time or episode of care.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 374 | 604
Participants | 95 | 72

4. Secondary Outcome: Number of Participants With Outpatient Hospital Visits After SARS-CoV-2 Infection
Description: In this outcome measure, number of participants with outpatient hospital visits who were fully vaccination and had SARS-CoV-2 breakthrough infection were analyzed. Outpatient hospital visits included an outpatient claim that occurs after the breakthrough COVID-19 diagnosis date or at the same time or episode of care other than emergency department visits.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 374 | 604
Participants | 146 | 164

5. Secondary Outcome: Number of Participants With Other Outpatient Visits After SARS-CoV-2 Infection
Description: In this outcome measure, number of participants with other outpatient visits (excluding emergency department visits and outpatient hospital visits) who were fully vaccination and had SARS-CoV-2 breakthrough infection were analyzed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 374 | 604
Participants | 309 | 527

6. Secondary Outcome: Number of Participants Hospitalized After SARS-CoV-2 Infection
Description: In this outcome measure, number of participants hospitalized who were fully vaccination and had SARS-CoV-2 breakthrough infection were analyzed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 374 | 604
Participants | 74 | 50

7. Secondary Outcome: Number of Participants Admitted to Intensive Care Unit (ICU) During Hospitalization After SARS-CoV-2 Infection
Description: In this outcome measure, number of participants admitted to ICU with or without Invasive Mechanical Ventilation (IMV) during hospitalization who were fully vaccination and had SARS-CoV-2 breakthrough infection were analyzed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 74 | 50
Participants
  With ICU admission and no IMV usage | 15 | 9
  With ICU admission and IMV usage | 8 | 1

8. Secondary Outcome: Number of Participants Who Received Invasive Mechanical Ventilation (IMV) During Hospitalization After SARS-CoV-2 Infection
Description: In this outcome measure, number of participants who received IMV with or without ICU admission during hospitalization who were fully vaccination and had SARS-CoV-2 breakthrough infection were analyzed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 74 | 50
Participants
  With ICU admission and IMV usage | 8 | 1
  No ICU admission with IMV usage | 1 | 0

9. Secondary Outcome: Number of Participants Died During Hospitalization After SARS-CoV-2 Infection
Description: In this outcome measure, number of participants who died during hospitalization who were fully vaccination and had SARS-CoV-2 breakthrough infection were analyzed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 74 | 50
Participants | 2 | 0

10. Secondary Outcome: Total Duration of Stay in Hospital After SARS-CoV-2 Infection
Description: Total duration of stay was total time spend by the participant for different types of hospitalization treatments, applicable for first hospitalization and/or readmissions.
Time Frame: From Dose 2 of COVID-19 vaccination till the end of study (retrospective data was retrieved and observed during 4 months of this study)
Population: Data was not collected and analyzed for this outcome measure as per Sponsor discretion.
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Total Expenditure on Healthcare Resource Utilization (HCRU) After SARS-CoV-2 Infection
Description: Total expenditure on HCRU was defined as total non-zero costs associated with any of the previously listed outpatient and inpatient encounters.
Time Frame: as for outcome 10
Population: Data was not collected and analyzed for this outcome measure as per Sponsor discretion.
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not planned to be collected hence time frame was not applicable
Description: In this study individual participant data was not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) cannot be met. Hence, AEs were not collected and reported in this study.
Arm/Group | BNT162b2 (Tozinameran): IC Cohort | BNT162b2 (Tozinameran): Non-IC Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data for outcome measures- Total duration of stay in hospital after SARS-COV-2 infection and total expenditure on healthcare resource utilization (HCRU) after SARS-COV-2 infection was not collected and analyzed as per Sponsor discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT05020145/Prot_SAP_000.pdf